CLINICAL TRIAL: NCT05038553
Title: CNS Pain Mechanisms in Early Rheumatoid Arthritis: Implications for the Acute to Chronic Pain Transition
Brief Title: Chronic Pain in Rheumatoid Arthritis
Acronym: CPIRA-2
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); University of Michigan (Other); Hospital for Special Surgery, New York (Other); University of Colorado, Denver (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Yvonne Lee, Associate Professor of Medicine and Preventive Medicine, Northwestern University
Other Study IDs: STU00211593; R01AR064850 (NIH)
Record Dates: First submitted 2021-08-30; First posted 2021-09-09 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Arthritis, Rheumatoid; Pain
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with early rheumatoid arthritis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The objective is to identify modifiable clinical factors and neurobiological pathways that lead to the development of chronic pain in patients with early rheumatoid arthritis. Participants will undergo quantitative sensory testing, a type of testing that involves assessing response to well-defined, quantifiable painful stimuli, at 0, 3, and 12 months. A subset of participants will also undergo magnetic resonance imaging at 0 and 12 months to assess neuroimaging markers that have previously been shown to be involved in chronic pain.

ELIGIBILITY:
Inclusion Criteria for QST:

1. Age ≥18 years
2. Meet either the 1987 or 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria for RA
3. Persistent joint symptoms ≤ 2 years
4. Active inflammatory disease
5. If taking opioids on an as needed (prn) basis, must be able to hold opioid for 12 hours before study procedures
6. If taking NSAIDs, must be able to hold NSAIDS for 24 hours before study procedures
7. If taking a central-acting pain medication, must be on a stable dose and able to stay on a stable dose throughout study

Exclusion Criteria for QST:

1. Routine, scheduled opioid use
2. Routine, scheduled prednisone dose >10 mg or its equivalent
3. Peripheral neuropathy
4. Peripheral vascular disease
5. Raynaud's phenomenon requiring treatment, manifested by claudication or ischemic rest pain
6. Uncontrolled blood pressure

Additional Inclusion Criteria for neuroimaging:

1. Age ≤ 80 years old
2. Right-handed or ambidextrous
3. Ability to lie on their back for the duration of the MRI scans

Additional Exclusion Criteria for neuroimaging:

1. Severe claustrophobia precluding MRI
2. Unable to fit comfortably in the MRI scanner (usually only occurs if body mass index >40 kg/m2)
3. Pregnant
4. Contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early RA recruited from academic medical centers
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia Survey Criteria | 12 months
  Minimum value 0, maximum value 31; higher scores indicate worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne C Lee, MD, MMSc, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - University of Colorado, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Hospital for Special Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: No